CLINICAL TRIAL: NCT04616859
Title: Combination of Alcohol and Energy Drinks in a Binge Drinking Pattern: Acute Effects and Gender Differences
Brief Title: Binge Drinking of Alcohol Mixed With Energy Drinks
Acronym: ENERGYBINGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HUGTP/ENERGYBINGE/PNSD/1; HUGTP/ENERGYBINGE/PNSD/1 (Other: Hospital Universitari Germans Trias i Pujol)
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Healthy; Alcohol Drinking
Keywords: alcohol binge drinking; alcohol; energy drinks; pharmacokinetics; caffeine; gender
MeSH Terms: conditions — Alcohol Drinking; Coitus | interventions — Ethanol; Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcohol and Energy Drink (AmED) (Experimental): The total volume of drink will be 761 ml in women and 969 ml in men. The doses will be divided into 6 fractions administered one every 15 min simulating a binge drinking pattern (80 min in total).
  Women: Ethanol 172 ml (55 g) + ED 589 ml Men: Ethanol 219 ml (70 g) + ED 750 ml
  Interventions: Dietary Supplement: Alcohol and Energy Drink (AmED)
- Alcohol and Energy drink Placebo (Active Comparator): The total volume of drink will be 761 ml in women and 969 ml in men. The doses will be divided into 6 fractions administered one every 15 min simulating a binge drinking pattern (80 min in total).
  Women: Ethanol 172 mL (55 g) + placebo ED (a non-caffeinated soft drink) 589 mL Men: Ethanol 219 mL(70 g) + placebo ED 750 mL (a non-caffeinated soft drink)
  Interventions: Dietary Supplement: Alcohol and Energy drink Placebo
- Alcohol placebo and Energy drink (Active Comparator): The total volume of drink will be 761 ml in women and 969 ml in men. The doses will be divided into 6 fractions administered one every 15 min simulating a binge drinking pattern (80 min in total).
  Women: Ethanol placebo (water) 172 mL + ED 589 mL Men: Ethanol placebo (water) 219 mL + ED 750 mL
  Interventions: Dietary Supplement: Alcohol placebo and Energy drink
- Alcohol placebo and Energy drink placebo (Placebo Comparator): The total volume of drink will be 761 ml in women and 969 ml in men. The doses will be divided into 6 fractions administered one every 15 min simulating a binge drinking pattern (80 min in total).
  Women: Ethanol placebo (water) 172 mL+ placebo ED (a non-caffeinated soft drink) 589 mL Men: Ethanol placebo (water) 219 mL + placebo ED (a non-caffeinated soft drinks) 750 mL
  Interventions: Dietary Supplement: Alcohol placebo and energy drink placebo

INTERVENTIONS:
Dietary Supplement: Alcohol and Energy Drink (AmED) — Multiple oral dose of alcohol mixed with ED
  Arms: Alcohol and Energy Drink (AmED)
Dietary Supplement: Alcohol and Energy drink Placebo — Multiple oral dose of alcohol mixed with ED placebo (soft drink)
  Arms: Alcohol and Energy drink Placebo
Dietary Supplement: Alcohol placebo and Energy drink — Multiple oral dose of alcohol placebo (water) mixed with ED
  Arms: Alcohol placebo and Energy drink
Dietary Supplement: Alcohol placebo and energy drink placebo — Multiple oral dose of alcohol placebo (water) mixed with ED placebo (soft drink)
  Arms: Alcohol placebo and Energy drink placebo

SUMMARY:
The purpose of the study is to assess the relevance of gender in the acute effects (subjective, physiological and driving-related skills) observed after controlled administration of alcohol in a binge-drinking pattern mixed with energy drinks (AmED)

DETAILED DESCRIPTION:
Consumption of alcohol mixed with energy drinks (AmED) has increased mainly among young people. Energy drinks (ED) are usually combined with alcohol with the intention of counteracting its effects. However, most studies have not shown a reduction in drunkenness and consumption is related with engagement of risk-taking behaviours like driving under alcohol effects. It is already known that alcohol concentrations and effects are higher in women than in men even after adjusting dose by weight.

The relevance of gender in the acute effects of alcohol associated with ED consumed in a binge-drinking pattern has been poorly studied. A randomized clinical trial will be conducted in healthy volunteers (1:1) and four treatment conditions will be administered: alcohol+ED, alcohol+placebo of ED, placebo of alcohol+ED and placebo of alcohol+placebo of ED. Subjective and physiological effects, driving related skills, and alcohol and caffeine concentrations will be measured along an 8-hours period. A pilot study has been conducted with the first 6 volunteers to select the alcohol doses. In the definitive study 70 g of alcohol in men and 55 g in women will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18-40 years old, weight between 50 and 100 kg and BMI (BMI=weight/height²) between 20-28 kg/m². Lower or higher BMIs will be allowed, if the researchers considered that do not suppose a risk to the subjects and do not interfere with the objectives of the study.
2. Recreational alcohol consumption in form of occasional binge-drinking (≥1 episode / month) and at least consumption of 1 unit (10 g, "standard" drink - one alcoholic drink equivalent) per day or its equivalent over the whole week [7 units, 70 g)]) and having experienced drunkenness several times
3. Regular consumption of beverages containing methylxanthines at least 7 per week (coffee, tea, chocolate, cola soda, energy drinks). Consumption of energy drinks at least once.
4. Understand and accept the study's procedures and sign an informed consent form.
5. No evidence of somatic or psychiatric disorders as per past medical history and physical examination.
6. The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.

Exclusion Criteria:

1. Not fill the inclusion criteria.
2. Pathological history or evidence of a preexisting condition (including gastrointestinal, liver, or kidney disorders) that may alter the absorption, distribution, metabolism or excretion of drugs or symptoms suggestive of drug-induced gastrointestinal irritation.
3. Present history of a substance use disorder according to Diagnostic and Statistical Manual for Mental Disorders (DSM-V), except for nicotine. Past history of mild substance use disorder (corresponding to substance abuse according to DSM-IV) could be included.
4. Previous or actual psychiatric disorders, alcoholism, abuse of prescription drugs or illegal substances or regular consumption of psychoactive drugs.
5. Having donated blood or having participated in this same study in the preceding 8 weeks, or having participated in any clinical trial with drugs in the preceding 12 weeks
6. Having had any somatic disease or having undergone major surgery in the 3 months prior to inclusion in the trial.
7. Individuals intolerant or having experienced a severe adverse reaction to alcohol or energy drinks. Asian subjects with no intolerance or no serious adverse reactions to alcohol could be included.
8. Having regularly taken medication in the month before the trial, except for vitamins, herb-based remedies, dietary supplements that if, according to the Principal Investigator or his appointed collaborators' opinion, they pose no threat to the subjects and they won't interfere with the study's objectives. Single doses of symptomatic drugs taken during the week before the experimental session will not constitute an exclusion criterion if it can be assumed that it has been completely eliminated on the day of the experimental session.
9. Smokers of >5 cigarettes/day
10. Consumption of >20 g/day of alcohol (females) or of >40 g/day (males)
11. Daily consumption of more than 5 coffees, teas, cola drinks or other stimulant or xanthine-containing beverages in the 3 months prior to inclusion in the study.
12. Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
13. Subjects with positive serology to Hepatitis B, C or HIV.
14. Pregnant, breastfeeding women and those using hormonal contraception,. Those not using an effective contraceptive (i.e. abstinence, intrauterine devices, barrier methods or partner vasectomy).
15. Women with amenorrhea or suffering severe premenstrual syndrome.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in subjective effects measured with Biphasic alcohol effects scale (BAES) | From baseline to 8 hours after administration
  Subjective effects of alcohol will be measured using Biphasic alcohol effects scale (0-70 points). Higher scores mean worse outcome. Obtained baseline and 1, 1.30, 2, 3, 4, 6 and 8-h after administration.
Change in psychomotor vigilance task (PVT) | From baseline to 6 hours after administration
  Test will be performed using a specific software. Mean latency will be measured. Obtained baseline and 1.30, 4 and 6-h after administration.

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC 0-8h) of ethanol blood concentrations | From baseline to 8 hours after administration
  Calculation of AUC of ethanol blood concentrations. Obtained baseline and 0.30h , 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Area under the concentration-time curve (AUC 0-8h) of ethanol breath concentrations | From baseline to 8 hours after administration
  Obtained baseline and 0.15, 0.30 , 0.45, 1, 1.15,1.30, 1.45, 2, 2.15, 2.30, 3, 4, 6 and 8-h after administration.
Area under the concentration-time curve (AUC 0-8h) of caffeine blood concentrations | From baseline to 8 hours after administration
  Calculation of AUC of caffeine concentrations obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Maximum concentration (Cmax) of ethanol in blood | From baseline to 8 hours after administration
  Maximum concentration (Cmax) of ethanol in blood
Maximum concentration (Cmax) of caffeine in plasma | From baseline to 8 hours after administration
  Maximum concentration (Cmax) of caffeine in plasma
Time to reach maximum concentration (tmax) of ethanol in blood | From baseline to 8 hours after administration
  Time to reach maximum concentration (tmax) of ethanol in blood
Time to reach maximum concentration (tmax) of ethanol in breath air | From baseline to 8 hours after administration
  Time to reach maximum concentration (tmax) of ethanol in breath air
Time to reach maximum concentration (tmax) of caffeine in plasma | From baseline to 8 hours after administration
  Time to reach maximum concentration (tmax) of caffeine in plasma
Area under the concentration-time curve (AUC 0-8h) of taurine plasma concentrations | From baseline to 8 hours after administration
  Calculation of AUC of taurine concentrations obtained baseline and 0.30h , 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration
Maximum concentration (Cmax) of taurine plasma concentrations | From baseline to 8 hours after administration
  Maximum concentration (Cmax) of taurine plasma concentrations
Time to reach maximum concentration (tmax) of taurine plasma concentrations | From baseline to 8 hours after administration
  Time to reach maximum concentration (tmax) of taurine plasma concentrations
Change in drunkenness feeling | From baseline to 8 hours after administration
  Drunkenness will be measured using a visual analog scale (0-100 mm). Higher scores mean worse outcome. Obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in dizziness feeling | From baseline to 8 hours after administration
  Dizziness will be measured using a visual analog scale (0-100 mm).Higher scores mean worse outcome. Obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in drowsiness feeling | From baseline to 8 hours after administration
  Drowsiness will be measured using a visual analog scale (0-100 mm). Higher scores mean worse outcome. Obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in palpitations reported by the participant | From baseline to 8 hours after administration
  Palpitations will be measured using a visual analog scale (0-100 mm). Higher scores mean worse outcome. Obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in anxiety feeling | From baseline to 8 hours after administration
  Anxiety will be measured using a visual analog scale (0-100 mm).Higher scores mean worse outcome. Obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in headache | From baseline to 8 hours after administration
  Headache will be measured using a visual analog scale (0-100 mm). Higher scores mean worse outcome. Obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in ability and predisposition to drive in certain situations | From baseline to 8 hours after administration
  Will be measured using a visual analog scale (0-100 mm).Higher scores mean worse outcome. Obtained baseline and 1.30, 4, 6 and 8-h after administration.
Desire to keep drinking | At 1.30 hours
  Will be measured using a visual analog scale (0-100 mm). Higher scores mean worse outcome. Obtained at the end of beverage administration. Only one measure at 1.30 hours.
Change in subjective effects measured with Addiction Research Center Inventory (ARCI) | From baseline to 8 hours after administration
  Obtained baseline and 1, 1.45, 4, 6 and 8-h after administration.
Change in blood pressure | From baseline to 8 hours after administration
  Systolic and diastolic blood pressure (mmHg) will be measured obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in heart rate | From baseline to 8 hours after administration
  Heart rate (beats/min) will be measured obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in oral temperature | From baseline to 8 hours after administration
  Oral temperature (ºC) will be measured obtained baseline and 0.30, 1, 1.30, 2, 2.30, 3, 4, 6 and 8-h after administration.
Change in Maddox Wing score (MW) | From baseline to 6 hours after administration
  Maddox wing is a device for the measurement of diopters of horizontal heterophoria. From 22 (exophoria) to 15 (esophoria). Higher scores mean worse outcome.Obtained baseline and 1.30, 4 and 6-h after administration.
Beverage identification | 8 hours after administration
  Beverage identification questionnaire.There is an option to select each treatment condition. Only measured at 8h after administration
Change in tracking test performance | From baseline to 6 hours after administration
  Test will be performed using a computer program. Total time outside the road and number of errors will be measured. Obtained baseline and 1.30, 4 and 6-h after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Pérez-Mañá, MD, PhD, Principal Investigator — Hospital Universitari Germans Trias i Pujol-IGTP
Locations (1):
- Hospital Universitari Germans Trias i Pujol-Institut d'Investigació en Ciències de la Salut Germans Trias i Pujol (IGTP), Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Hladun O, Papaseit E, Poyatos L, Martin S, Perez-Acevedo AP, Barriocanal AM, Bustos-Cardona T, Malumbres S, De La Torre R, Langohr K, Farre M, Perez-Mana C. No significant gender differences in driving-related skills following alcohol mixed with energy drinks during an experimental binge-drinking episode. Front Pharmacol. 2025 May 23;16:1581229. doi: 10.3389/fphar.2025.1581229. eCollection 2025. PMID 40487410